CLINICAL TRIAL: NCT05933954
Title: Double-blind Randomized Controlled Study of the Effects of 5G Radiation on Skin
Brief Title: The Effects of 5G Radiation on Skin
Acronym: SEAwave
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Olivier Gaide, MD-PhD (Other)
Responsible Party: Sponsor-Investigator, Prof. Olivier Gaide, MD-PhD, Associate Professor, Médecin Chef, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CHUV-DD-00884-SEAWAVE-2023
Record Dates: First submitted 2023-06-19; First posted 2023-07-06 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Electromagnetic Radiation (5GFR2)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computer assisted randomisation of exposure vs non exposure side
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteers 5G-FR2 exposed vs sham-exposed skin (Other): A 5G source, only exposing a small skin-area, will be placed on each arm of the participants. Only one of the two sources will emit waves (controlled by a computer). One arm will be exposed to 20W/m2 (a dose rate inferior to the recommended maximum for EMW exposure in Switzerland), the other not (sham-exposed). The exposure time is 20 min.
  Interventions: Radiation: 5GFR2 non ionizing EMW exposure
- Patients with dermatoporosis 5G-FR2 exposed vs sham-exposed skin (Other): A 5G source, only exposing a small skin-area, will be placed on each arm of the participants. Only one of the two sources will emit waves (controlled by a computer). One arm will be exposed to 20W/m2 (a dose rate inferior to the recommended maximum for EMW exposure in Switzerland), the other not (sham-exposed). The exposure time is 20 min.
  Interventions: Radiation: 5GFR2 non ionizing EMW exposure
- Patients with atopic dermatitis 5G-FR2 exposed vs sham-exposed skin (Other): A 5G source, only exposing a small skin-area, will be placed on each arm of the participants. Only one of the two sources will emit waves (controlled by a computer). One arm will be exposed to 20W/m2 (a dose rate inferior to the recommended maximum for EMW exposure in Switzerland), the other not (sham-exposed). The exposure time is 20 min.
  Interventions: Radiation: 5GFR2 non ionizing EMW exposure
- Skin-cancer prone patients 5G-FR2 exposed vs sham-exposed skin (Other): A 5G source, only exposing a small skin-area, will be placed on each arm of the participants. Only one of the two sources will emit waves (controlled by a computer). One arm will be exposed to 20W/m2 (a dose rate inferior to the recommended maximum for EMW exposure in Switzerland), the other not (sham-exposed). The exposure time is 20 min.
  Interventions: Radiation: 5GFR2 non ionizing EMW exposure

INTERVENTIONS:
Radiation: 5GFR2 non ionizing EMW exposure — A 5G source, only exposing a small skin-area, will be placed on each arm of the participants. Only one of the two sources will emit waves (controlled by a computer). One arm will be exposed to 20W/m2 (a dose rate inferior to the recommended maximum for EMW exposure in Switzerland), the other not. The exposure time is 20 minutes.
  After the exposure, the participants will wait one hour and a 7.5-mm biopsy by punch (two pieces: one 5-mm punch + half a 5-mm punch) will be performed under local anesthesia on each arm. The wound will be closed by a simple suture. A second set of samples will be taken 24h after the exposure, using the same procedure.
  For each participant, 1 full biopsy per arm and per time-point will be used for single-cell-RNA-sequencing analysis. The selected method uses generic probed sequencing and does not generate patient-specific genomic information.

SUMMARY:
The current 5G waves used on the daily life are ranging from 410 MHz to 7125 MHz and are called FR1. The next deployed 5G waves will be FR2, from 24.45 GHz to 52.6 GHz. Our project targets the 27.5 GHz frequency, as it will be used in both Europe and the USA. Recent studies have shown that these 5G FR2 waves enter the skin but do not penetrate deeper in the body, which is why our project focuses on the skin.

Our aim is to understand the effects of 5G waves on skin by performing a clinical trial. In this study, participants (healthy volunteers, patients with dermatoporosis, or whose skin is prone to developing cancer or who suffer from atopic dermatitis) will be exposed to carefully chosen 5G parameters and skin will be analyzed by state-of-the-art single cell RNA analysis (an unbiased and very sensitive technique ideal for studying cell behavior changes). This project will also decipher the differences between women and men, in response to 5G FR2 waves.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited in accordance with European and Swiss standards for the following groups: Healtyh volunteers or Dermatoporosis defined as a chronic skin fragility syndrome orGorlin Goltz Syndrome defined as OMIM 10940014, or Familial Cylindromatosis or SB Syndrome defined as OMIM 132700/60504114, or XPV defined as OMIM 27875014 or Atopic dermatitis defined as a chronic inflammatory skin disease characterised by eczematous skin lesions and intense pruritus
* Able to give informed consent as documented by signature,
* Adults, from 18 to 80 yo, according to groups

Exclusion Criteria:

* Recent intense exposure to sun (defined as causing a sunburn, within the last 7 days)
* Pregnant (excluded with a pregnancy test) or lactating women,
* Patients taking anti-coagulants
* Clinically significant concomitant diseases (cutaneous exam by the specialist),
* Active enrolment in another clinical trial,
* Participants incapable of judgment or participants under tutelage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Variation in expression levels of proteins expressed by skin cells, comparing exposed and non-exposed skin | 18 month
  Measure: Fold of expression of messenger RNAs, as measured by single cell RNA analysis. This is measure of the overall tissue composition and cellular activity.
  Further information:
  Inputs: ScRNAseq data from the sample, age, sex, groups, skin thickness, arm of the biopsy, 1h or 24h after exposure, concomitant medication, healing process, adverse effects.
  Outputs: based on our own analyses and others (ref). We will use Seurat package to perfom the quality controls of the data on individual samples, then integrate the samples for each patient to analyze their inter-variability. To determine cell types, we will combine unsupervised clustering and differential expression to compare top differentially expressed genes (using Wilcoxon rank sum tests of the FindMarker function of Seurat) with cell type specific expression known from literature. We will also use ProjecTILs package30 to define more precisely the immune subtypes.

SECONDARY OUTCOMES:
Variation in expression levels of proteins expressed by skin cells, comparing female and male skin | 18 month
  Measure: Fold of expression of messenger RNAs, as measured by single cell RNA analysis. This is measure of the overall tissue composition and cellular activity. For further details, see primary outcome.
Variation in expression levels of proteins expressed by skin cells, comparing healthy skin and disease-affected skin | 18 month
  Measure: Fold of expression of messenger RNAs, as measured by single cell RNA analysis. This is measure of the overall tissue composition and cellular activity. For further details, see primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pich-Bavastro C, Yerly L, Di Domizio J, Tissot-Renaud S, Gilliet M, Kuonen F. Activin A-Mediated Polarization of Cancer-Associated Fibroblasts and Macrophages Confers Resistance to Checkpoint Immunotherapy in Skin Cancer. Clin Cancer Res. 2023 Sep 1;29(17):3498-3513. doi: 10.1158/1078-0432.CCR-23-0219. PMID 37327314